CLINICAL TRIAL: NCT00603681
Title: Non-Inferiority Study; Comparison of Polyethylene Glycol Solution With and Without Electrolytes for Treatment of Chronic Constipation in Elderly Institutionalised Patients: a Double-Blind, Randomised, Parallel-Group, Multicentre Study
Brief Title: Comparison of PEG Solutions With and Without Electrolytes in the Treatment of Constipation
Acronym: PEGorion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Ulla Sairanen, Orion Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3066001
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Constipation
Keywords: constipation; aged; polyethylene glycol
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 4000; Electrolytes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T (Experimental): Test product
  Interventions: Drug: Polyethylene glycol 4000
- C (Active Comparator): Reference product
  Interventions: Drug: Polyethylene glycol 4000 with electrolytes

INTERVENTIONS:
Drug: Polyethylene glycol 4000 — powder for oral solution 12 g of PEG once a day, twice a day or once every other day for 4 weeks
  Other Names: Pegorion
  Arms: T
Drug: Polyethylene glycol 4000 with electrolytes — granules for oral solution 12 g of PEG once a day, twice a day or once every other day for 4 weeks
  Other Names: Colonsoft
  Arms: C

SUMMARY:
The aim of the study is to show that new polyethylene glycol (PEG) solution without electrolytes is as effective in the treatment of constipation as PEG solution with electrolytes in the elderly institutionalized people. Also, the tolerability and the safety of the study drug will be examined.

DETAILED DESCRIPTION:
Constipation is a major problem in elderly institutionalised patients. Non-pharmacological treatments are proposed as primary management of constipation, but institutionalised patients are not likely to be able to increase either the intake of dietary fibre or fluid and their physical activity is low.

The latest agent widely used for the treatment of constipation is polyethylene glycol (PEG). PEG is classified into the group of osmotic laxatives. It is minimally absorbed from the gastrointestinal tract and not metabolised by colonic bacteria.

Most of the PEG products at the market contain electrolytes and have a salty and unpleasant taste which may affect the compliance of using them. A PEG solution without electrolytes has been developed and used for some years in various countries. Now we will compare the efficacy and safety of PEG solutions with or without electrolytes and their acceptability in the use for constipation in institutionalised patients.

ELIGIBILITY:
Inclusion Criteria:

* Isotonic PEG treatment for constipation at the stable dose for at least 2 weeks before the run-in period

Exclusion Criteria:

* Other medical treatment for constipation than isotonic PEG or plantago ovata seeds
* Severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Stool frequency | week 4

SECONDARY OUTCOMES:
Stool frequency | Week 2
Stool straining | Weeks 2 and 4
Stool consistency | Weeks 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Seinelä, MD, Principal Investigator — Pirkanmaan erikoislääkäripalvelu Oy; Ulla Sairanen, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (10):
- Finland (10):
  - Koskikoti, Tampere
  - Koivupirtti, Tampere
  - Tampereen sotainvalidien Veljeskoti, Tampere
  - Lahdensivun koti, Tampere
  - Nurmikoti, Tampere
  - Vire Koti Kaukaharju assisted-living facility, Tampere
  - Taatala assested-living facility, Tampere
  - Kuusela assisted-living facility, Tampere
  - Petäjäkoti, Tampere
  - Nursing home of Tiuravuori, Ylöjärvi